CLINICAL TRIAL: NCT00929058
Title: Bevacizumab and Vasoconstriction
Acronym: BVZ1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Paul Smits, UMCN
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BVZ1
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2009-06

CONDITIONS: Hypertension; Cancer
MeSH Terms: conditions — Hypertension; Neoplasms | interventions — Bevacizumab

ARMS (1):
- Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Intra-arterial infusion during 6 minutes

SUMMARY:
Rationale: The introduction of angiogenesis inhibitors has remarkably improved treatment of patients with several types of cancer. One of the most common side effects of angiogenesis inhibitors is hypertension. In patients treated with bevacizumab hypertension had an overall incidence up to 32%. The etiology of hypertension caused by treatment with angiogenesis inhibitors is unclear.

Objective: To study if arterial bevacizumab infusion causes acute vasoconstriction using plethysmography in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male 18-50 years old
* normal results of glucose, lipids and creatinine
* informed consent

Exclusion Criteria:

* History of abuse of drugs or alcohol
* History of malignant disease
* First degree relatives with a history of cancer before the age of 50
* First degree relatives with a history of premature cardiovascular disease
* Current use of medication
* Clinical evidence of cardiac of pulmonary disease
* Hypertension ( systolic>140mmHg, diastolic >90mmHg)
* Diabetes mellitus
* smoking
* a history of thombosis or a family history of recurrent thrombosis
* abnormality on ECG

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Fore-arm vasomotor response to administered bevacizumab, expressed as percentage change in forearm blood flow ratio | Infusion of bevacizumab during 6 minutes

SECONDARY OUTCOMES:
Correlation between VEGF concentrations in plasma and the vasoconstrictive response to bevacizumab | Infusion of bevacizumab during 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD PhD, Principal Investigator — UMCN
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands